CLINICAL TRIAL: NCT00006013
Title: Phase II Trial of SU5416 as Treatment for Refractory/Relapsed Multiple Myeloma
Brief Title: SU5416 in Treating Patients With Refractory or Relapsed Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FCCC-00009; CDR0000068022 (Registry Identifier: PDQ (Physician Data Query)); NCI-58 (Other Grant/Funding Number: NCI)
Record Dates: First submitted 2000-07-05; First posted 2003-06-25 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Semaxinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: semaxanib

SUMMARY:
RATIONALE: SU5416 may stop the growth of multiple myeloma by stopping blood flow to the cancer cells.

PURPOSE: Phase II trial to study the effectiveness of SU5416 in treating patients who have refractory or relapsed multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate and response duration of patients with refractory or relapsed multiple myeloma treated with SU5416. II. Determine the toxicity of SU5416 in this patient population.

OUTLINE: This is a multicenter study. Patients receive SU5416 IV over 1 hour twice weekly. Treatment continues in the absence of unacceptable toxicity or disease progression. Patients are followed for survival.

PROJECTED ACCRUAL: A total of 20-38 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed multiple myeloma with an elevated monoclonal protein in serum and/or urine No history of CNS lesion or CNS bleed

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Cytopenias secondary to multiple myeloma involvement of bone marrow allowed Cytopenias not due to multiple myeloma require: WBC at least 3,000/mm3 Platelet count at least 75,000/mm3 Hepatic: Transaminases no greater than 2 times upper limit of normal Bilirubin no greater than 1.5 mg/dL Renal: Creatinine no greater than 2.0 mg/dL OR Creatinine clearance at least 50 mL/min Cardiovascular: No congestive heart failure, severe peripheral vascular disease, or significant arrhythmia No poorly controlled systolic or diastolic hypertension No uncompensated coronary artery disease No history of myocardial infarction or severe/unstable angina within past 6 months No known hypercoagulable state or deep venous or arterial thrombosis within past 3 months Pulmonary: No pulmonary embolism within past 3 months Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 3 months after study No other severe medical or psychiatric condition (e.g., active peptic ulcer, active infection, or history of severe alcohol or drug abuse) No known hypersensitivity to paclitaxel or Cremophor

PRIOR CONCURRENT THERAPY: Biologic therapy: See Chemotherapy Chemotherapy: At least 1 but no more than 3 prior chemotherapy regimens Induction followed by high dose therapy with stem cell support considered a single treatment regimen Tandem courses of high dose therapy considered as 2 regimens Endocrine therapy: At least 1 prior regimen containing steroids Radiotherapy: Prior radiotherapy for symptom control allowed Surgery: At least 3 weeks since prior major surgery At least 1 year since prior coronary artery surgery, angioplasty, or stent placement No prior brain surgery Other: No other concurrent investigational drugs Concurrent bisphosphonates (e.g., pamidronate) allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2000-06; Primary Completion 2003-01 (Actual); Study Completion 2003-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell R. Smith, MD, PhD, Study Chair — Fox Chase Cancer Center
Locations (4):
- United States (4):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee